CLINICAL TRIAL: NCT03893968
Title: Are Doctors and Assistant Nurses Equally Good at Informing Patients: A Randomized Controlled Trial Comparing Information Recall Regarding Postoperative Self-care
Brief Title: Are Doctors and Assistant Nurses Equally Good at Informing Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, Aleksandra McGrath, Senior Consultant, Umeå University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2017/446-31
Record Dates: First submitted 2018-12-17; First posted 2019-03-28 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Patient Care

STUDY DESIGN:
Intervention Model Description: Patients are assigned to either a group informed by doctors or assistance nurses in parallel.
Who Masked: Investigator
Masking Description: The investigator is blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Informed by a doctor (Experimental): Information by a doctor
  Interventions: Behavioral: Information by a doctor
- Informed by an assistant nurse (Experimental): Information by an assistant nurse
  Interventions: Behavioral: Information by an assistant nurse

INTERVENTIONS:
Behavioral: Information by an assistant nurse — Information received by patients after ambulatory hand surgery under local anaesthetic about postoperative self care given by an assistent nurse.
  Arms: Informed by an assistant nurse
Behavioral: Information by a doctor — Information received by patients after ambulatory hand surgery under local anaesthetic about postoperative self care given by a doctor.
  Arms: Informed by a doctor

SUMMARY:
Objectives: to compare patients' recall of information regarding postoperative self-care when being informed by either doctors or assistant nurses.

Methods: a non-blinded randomized single-center controlled trial being conducted at a hand-surgical unit in Northern Sweden. Included are adult ambulatory patients about to undergo surgery in local anesthesia. Patients are randomized into two parallel groups, with the control-group being informed by doctors and the intervention-group by assistant nurses. Patients will be telephoned one week after surgery for assessment of information recall via a structured telephone-interview.

DETAILED DESCRIPTION:
The study was conducted within the hand-surgical unit at Norrland's University Hospital in Umeå, county of Västerbotten, in Sweden. There are three hospitals in this sparsely populated county of 55432〖km〗^2 with about 268000 in population. The hand-surgery unit serves both the local population and is a tertiary referral center.

As the healthcare in Sweden is funded by taxpayers, the healthcare for patients is free, apart from a small nominal fee. There was a total of seven doctors and seven assistant nurses participating in the study, all having several years of experience working with hand-surgical care. Prior to the study, doctors had the formal responsibility of informing patients about their postoperative care. However, despite it being the surgeons' responsibility, the task of informing patients was at times performed by assistant nurses. After receiving the information, patients were discharged and left the clinic. Normally patients receive a complementary written information after being informed verbally. Patients included in the study did not receive the written information, since it might have been a confounding factor in understanding of information.

ELIGIBILITY:
Inclusion Criteria:

* about to undergo elective hand surgical procedure in local anaesthesia
* 18 years or older.

Exclusion Criteria:

* does not speak Swedish
* dementia or other form av cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Information recall | 1 week after surgery
  A telephone-interviews were performed seven days after the surgery using a structured questionnaire. For the main objective, seven questions were asked testing patients recall/knowledge of their postoperative self-care. Each question evaluated the patients' knowledge of a unique aspect of postoperative self-care. The questionnaire is designed based on the postoperative info sheet received by patients after hand surgery.

SECONDARY OUTCOMES:
Stress and satisfaction | 1 week after surgery
  During the telephone interview the patients could rate on a 1-10 scale their level of "feeling of understood the information", stress, and satisfaction. "Feeling of having understood the information" means the patients perception of having fully understood all the information and knowing fully what to do when leaving the hospital. For assessing "stress", the interviewer asked about the level of stress that the patient had experienced during the week following the surgery. Regarding "satisfaction", the interviewer asked and assessed how satisfied the patients were with the way the personnel had informed the patient (e.g. not used difficult or confusing language, had given the patient time to ask questions etc).
Additional healthcare contacts | 30 days after surgery
  Compare differences in the number of healthcare contacts due to not being able to recall or having understood information.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Fahlström, Study Chair — Umea University
Locations (1):
- Norrland's University Hospital, Umeå, Sverige, Sweden

IPD SHARING:
Plan to Share IPD: No